CLINICAL TRIAL: NCT03121339
Title: A Phase 1, Open-Label, Randomized, 2×2 Crossover Study of Pharmacodynamics Comparing the Impact of Tablet Size and Fasting Status With an Oral Human Influenza A/California/04/2009 (H1N1) HA Adenoviral-Vector Based Vaccine and dsRNA Adjuvant
Brief Title: Pharmacodynamic Open-Label Trial With VXA-A1.1 Oral H1 Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VXA02-RLT-01
Record Dates: First submitted 2017-04-14; First posted 2017-04-20 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Seasonal Influenza Preventative Vaccine Pharmacodynamics

STUDY DESIGN:
Intervention Model Description: open-label with two tablet sizes labeled with different radioisotopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A - Fasting Condition (Active Comparator): Radio-labeled VXA-A1.1 H1 Tablet Vaccine (small) and VXA-A1.1 H1 Tablet Vaccine (large) will be administered to fasted subjects.
  Interventions: Biological: VXA-A1.1 H1 Tablet Vaccine (small); Biological: VXA-A1.1 H1 Tablet Vaccine (large)
- Treatment B - Fed Condition (Active Comparator): Radio-labeled VXA-A1.1 H1 Tablet Vaccine (small) and VXA-A1.1 H1 Tablet Vaccine (large) will be administered to subjects with a small snack.
  Interventions: Biological: VXA-A1.1 H1 Tablet Vaccine (small); Biological: VXA-A1.1 H1 Tablet Vaccine (large)

INTERVENTIONS:
Biological: VXA-A1.1 H1 Tablet Vaccine (small) — Tableted oral H1 vaccine (~140 mg tablet)
Biological: VXA-A1.1 H1 Tablet Vaccine (large) — Tableted oral H1 vaccine (~275 mg tablet)

SUMMARY:
This is a phase 1 open-label pharmacodynamics study in healthy adults. The purpose of the study is to determine if the tablet formulation size of VXA-A1.1, an adjuvanted adenoviral based influenza vaccine, has an impact on delivery location. The secondary objective is to evaluate delivery with fasting versus fed status.

DETAILED DESCRIPTION:
This is a pharmacodynamics study in healthy adult males. The purpose of the study is to determine if the tablet formulation size of VXA-A1.1, an adjuvanted adenoviral based influenza vaccine, impacts the location and time of initial and complete disintegration of the drug product. The secondary objective is to evaluate delivery with fasting versus fed status.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers aged 18 - 49 years, inclusive
* Willing and able to give written informed consent/HIPAA authorization form
* In good health (no clinically significant health concerns), as determined by medical history, physical examination, 12-lead ECG, vital signs and laboratory tests at screening
* Liver function tests (alanine aminotransferase (ALT), aspartate amino transferase (AST), alkaline phosphatase (ALP), direct bilirubin (DB) and total bilirubin (TB) are within the normal range. [N.B., an elevated TB in the absence of an elevated direct bilirubin (benign unconjugated hyperbilirubinemia, known as Gilbert's Syndrome) will not be exclusionary]
* Body weight ≥ 50 kg and a Body mass index between 17 and 35 at screening
* Willingness to abstain from caffeine or xanthine containing foods or beverages, alcohol, tobacco or nicotine-containing products and strenuous exercise from 72 hours prior to screening and each dosing until discharge post each Dosing Day.
* Dietary habits that fall within the range of normal, as determined by the Investigator. Examples of abnormal diets are liquid diets, protein only diets, high fat diets, or low carbohydrate diets.
* Verbal confirmation from subject that his bowel movements are regular.
* Comprehension of the study requirements (in English) with ability and willingness to complete all assessments and comply with scheduled visits and contacts.

Exclusion Criteria:

* Administration of any vaccine within 4 weeks preceding DP administration or during the study through the active period (Day 36), or any licensed or investigational adjuvanted vaccine within 12 months preceding DP administration, or planned use of any licensed or investigational adjuvanted vaccine during the study through the 12-month safety follow- up period
* Use of any investigational drug or device the greater of: within 4 weeks preceding DP administration, or planned use of the above stated during the study through the study active period (Day 36) OR within 5 half-lives of an investigational drug product
* Use of concomitant medications that may interfere with normal gastrointestinal tract function, including but not limited to those listed below:

  1. Proton pump inhibitors
  2. H2 blockers
  3. GI motility stimulants (e.g. metoclopramide)
  4. Anti-nausea/anti-emetics
  5. Opiate class pain relievers
  6. Anti-diarrheals
  7. Laxatives
* Presence of significant uncontrolled medical or psychiatric illness (acute or chronic) including institution of new medical/surgical treatment or significant dose alteration for uncontrolled symptoms or drug toxicity within 3 months of screening
* Any one of the following ECG findings within 30 days prior to administration:

  1. QTc F (interval duration > 450 msec (male),
  2. QRS interval greater than 120 msec,
  3. PR interval greater than 220 msec,
  4. Clinically significant ST-T wave changes or pathologic Q waves
* Positive serology for HIV-1 or HIV-2, or HBsAg or HCV antibodies
* Cancer, or treatment for cancer, within past 3 years (excluding basal cell carcinoma, squamous cell carcinoma, and cervical cancer in situ)
* Radiation exposure from clinical trials, including that from the present study, and from diagnostic X-rays, but excluding background radiation, exceeding a target organ (colon) dose of 50 mSv (5 rems) from a single dose within the last 30 days or a cumulative dose of 150 mSv (15 rems) in the last 12 months. No subject whose occupation requires monitoring for radiation exposure may be enrolled in the study.
* Presence of household members who are neonates, pregnant women, or hematopoietic stem cell transplant or solid organ transplant recipients or who are immunocompromised including those who are HIV positive.
* History of drug, alcohol or chemical abuse within 1 year prior to administration
* Acute disease within 72 hours prior to administration defined as the presence of a moderate or severe illness with or without fever (as determined by the Investigator through medical history and physical examination) or any acute respiratory or gastrointestinal illness even with mild symptoms occurring within 7 days of administration
* Presence of a fever ≥ 38ºC measured orally at baseline
* Positive urine drug screen for drugs of abuse at screening
* Positive breath or urine alcohol test at screening
* Consistent/habitual smoking (> 10 cigarettes/day) within 6 months prior to administration
* History or presence of acute/chronic diarrhea or constipation
* History of serious reactions to any vaccination such as anaphylaxis, respiratory problems, Guillain-Barre syndrome, hives or abdominal pain
* History of a hypersensitivity or allergic reaction to any component of the investigational DP, including but not limited to fish gelatin
* History of irritable bowel disease or inflammatory digestive or gastrointestinal condition that could affect the distribution / safety evaluation of an orally administered DP targeting the mucosa of the small intestine. Such conditions may include but are not limited to:

  1. Esophageal Motility Disorder
  2. Malignancy
  3. Malabsorption
  4. Pancreaticobiliary disorders
  5. Irritable bowel syndrome
  6. Celiac Disease
  7. Inflammatory Bowel Disease
  8. Surgical Resection with the exception of appendectomy or a minor resection that is deemed acceptable by investigator and sponsor
  9. GERD
  10. Hiatal Hernia
  11. Peptic Ulcer (History of cholecystectomy is not exclusionary)
* Any condition that resulted in the absence or removal of the spleen
* History of any form of angioedema
* Male subject who is unwilling to use an acceptable method of contraception, as listed below, for the duration of the study and continuing for 90 days after the subject's last study DP dose. Acceptable methods of contraception include the following: (1) complete abstinence from intercourse beginning with the first dose of study DP and continuing for 90 days after the final study DP dose, (2) male subject sterilization (vasectomy), (3) sterilization of or non-childbearing potential female partner (bilateral tubal ligation/salpingectomy, hysterectomy, post-menopausal), (4) use of hormonal contraception by female partner (implantable, patch, oral, injectable), (5) use of an intrauterine device (IUD) or intrauterine system by female partner, (6) barrier methods (condom by male or an occlusive cap [diaphragm or cervical/vault caps] by female partner) with concomitant spermicidal foam/gel/film/cream/suppository use, (7) any other birth control method with published data showing a failure rate that is < 1% per year. Male subjects should not donate sperm for the duration of the study and for 90 days after the last DP dose. Male subjects who are not sexually active but become active, must comply with the contraceptive requirements above.
* Any condition that, in the opinion of the Investigator, might interfere with ability to assess the primary study objectives

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2018-04-03 (Actual)

PRIMARY OUTCOMES:
PD: Location of disintegration | 7 days
  Site of initial and complete disintegration of the study DP
PD: Time to disintegration | 7 days
  Time of initial and complete disintegration of the study DP

CONTACTS AND LOCATIONS:
Overall Officials: David Liebowitz, MD, PhD, Study Director — Vaxart, Inc.
Locations (1):
- Scintipharma, Inc., Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No